CLINICAL TRIAL: NCT04772222
Title: Dexmedetomidine Use in Infants Undergoing Cooling Due to Neonatal Encephalopathy (DICE Trial)
Acronym: DICE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Mariana Baserga, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 136561
Record Dates: First submitted 2021-02-18; First posted 2021-02-26 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Pain
Keywords: Therapeutic hypothermia; dexmedetomidine
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Pain | interventions — Dexmedetomidine; Morphine

STUDY DESIGN:
Intervention Model Description: Infants randomized to receive open-label dexmedetomidine (DMT) or morphine for pain and sedation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (DMT) (Experimental): Subjects randomized to DMT arm in a 1:1 ratio. A loading dose of 1 mcg/kg will be given followed by 0.1 to 0.5 mcg/kg/h continuous infusion. The Neonatal Pain, Agitation, and Sedation Scale (N-PASS) will be used to determine infusion rate.
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Morphine (Active Comparator): Subjects randomized to morphine in a 1:1 ratio. Intermittent dosing every 3-4 hours of 0.02-0.05 mg/kg/dose or continuous infusion of 0.005 to 0.01 mg/kg/hr. The N-PASS will be used to determine dosing and frequency.
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Potent α2-adrenergic receptor agonist that provides sedation, analgesia, and prevents shivering but does not suppress ventilation.
  Arms: Dexmedetomidine (DMT)
Drug: Morphine Sulfate — Opioid agonist that provides analgesia, pain management and sedation and may suppress ventilation.
  Arms: Morphine

SUMMARY:
Management of neonatal pain and sedation often includes opioid therapy. A growing body of evidence suggests long-term harm associated with neonatal opioid exposure. Providing optimal sedation while neonates are undergoing therapeutic hypothermia (TH) may be beneficial but also presents therapeutic challenges. While there is evidence from animal models of brain injury and clinical trials in adults to support the safety and neuroprotective properties of dexmedetomidine (DMT), there are no published large clinical trials demonstrating safety and efficacy of DMT use in neonates with hypoxic-ischemic encephalopathy (HIE) during treatment with TH. This study is innovative in proposing a Phase II, 2-arm trial providing the opportunity to evaluate the use of DMT as compared to the use of morphine for sedation and pain management for babies undergoing TH. We propose to confirm optimal DMT dosing by collecting opportunistic pharmacokinetics (PK) data and determine safety of DMT in this population. These data will inform a larger phase III efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Neonates ≥36 weeks' gestational age diagnosed with moderate-to-severe neonatal encephalopathy and treated with TH (target temperature 33.5°C) for a planned duration of 72 h.
* Infants requiring sedation and/or treatment to prevent shivering during TH as assessed by the Neonatal Pain, Agitation, and Sedation Scale (N-PASS) scores and a modified Bedside Shivering Assessment Scale.
* Informed consent document approved by the Institutional Review Board (IRB) obtained prior to randomization

Exclusion Criteria:

* Known chromosomal anomalies
* Cyanotic congenital heart defects
* Redirection of care being considered because of moribund condition, or a decision made to withhold full support

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Examine Safety Measures in infants receiving DMT to those receiving morphine | First 96 hours of life
  Safety will be evaluated during the first 4 days of life by documenting potential adverse events such hypotension, hypertension, bradycardia, cardiac arrhythmias, hypothermia, acute renal failure, liver failure, and seizures outside of normal range for the study population.

SECONDARY OUTCOMES:
DMT plasma levels | one week
  Two opportunistic PK samples (at time of routine laboratories) and a PK sample any time there is an adverse event will be obtained for measurement of DMT plasma concentrations as needed.

OTHER OUTCOMES:
Number of participants who experience shivering | First 96 hours of life
  Number of babies who experience shivering during therapeutic hypothermia will be compared between the two drug treatment regimens
Number of participants who require respiratory support | First week of life
  Number of babies who require respiratory support will be compared between the two drug treatment regimens. This will include ventilator, continuous positive airway pressure, and oxygen use
Days to full oral feedings by bottle or breast | Up to two months
  Days to full oral feedings will be compared between the two drug treatment regimens
Generalized Motor Assessment Scores (GMA) 7 days after weaned off of study drug or discharge, whichever happens first | up to 3 weeks
  the GMA is a validated test that aids in early detection of neurological movement disorders by evaluating the quality of movements during a 2-minute video. Certified assessors will grade the quality of movements which include: normal writhing, poor repertoire, cramped synchronized, and chaotic movements. All movements other than normal writhing are considered atypical. The results will be compared between the two drug treatments.
Generalized Motor Assessment Scores at 3-4 months of age | 3-4 months of age
  the GMA is a validated test that aids in early detection of neurological movement disorders by evaluating the quality of movements during a 2-minute video. Certified assessors will grade the quality of movements which include: normal writhing, poor repertoire, cramped synchronized, and chaotic movements. All movements other than normal writhing are considered atypical. The results will be compared between the two drug treatments.
Hammersmith Infant Neurological Exam (HINE) scores at 3-4 months of age | 3-4 months of age
  The HINE is a 26 item exam that assesses different aspects of neurological function and these scores will be compared between the two drug treatment regimens. This assessment scores 5 different neurological development areas: Cranial nerve function, posture, movements, tone, and reflexes/reactions. The maximum score is 78 and lowest score is 0. Higher scores show better neurological development consistent with better outcomes.
Hammersmith Infant Neurological Exam (HINE) scores at 6-9 months of age | 6-9 months of age
  The HINE is a 26 item exam that assesses different aspects of neurological function and these scores will be compared between the two drug treatment regimens. This assessment scores 5 different neurological development areas: Cranial nerve function, posture, movements, tone, and reflexes/reactions. The maximum score is 78 and lowest score is 0. Higher scores show better neurological development consistent with better outcomes.
Test of Infant Motor Performance (TIMP) scores at 3-4 months of corrected age | 3-4 months of corrected age
  This test evaluates posture and motor control and is designed to be used specifically in infants born prematurely. Results are given based on z-scores from normative values and are given as low average, below average, and far below average. Lower scores are more predictive of worse outcomes. These scores will be compared between the two drug treatment regimens.
Peabody Developmental Motor Skills (PDMS-2) at 6-9 months of age | 6-9 months of age
  This test evaluates fine motor, gross motor, and total motor skills. Results are converted to age equivalent rating and then quotient scores are given for each category. Minimum is 35 and maximum is 165. The average score is 90-110, with higher scores given in 3 SD above average performance and lower scores given in 3 SD below average performance.The higher the score, the better predicted outcome. These scores will be compared between the two drug treatment regimens.
Ages and Stages Questionnaire at 6-9 months of age | 6-9 months of age
  Parental survey that assesses communication, gross and fine motor skills, and social behaviors. Scores range from 0-60, and the higher the score, the better the outcome.
  These scores will be compared between the two drug treatment regimens

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Baserga, MD, Principal Investigator — University of Utah
Locations (5):
- United States (5):
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley Hospital, Provo, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Utah Health, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No